CLINICAL TRIAL: NCT06251310
Title: A Phase 1a/1b Dose Escalation, Dose Expansion Study of SW-682 in Participants With Advanced Solid Tumors Enriched for Those With Hippo Pathway Mutations
Brief Title: SW-682 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TEAD-AST-101
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Mesothelioma, Malignant
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two sequential parts: Part 1 dose escalation and Part 2 dose expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 Dose Escalation Cohorts Ranging in Dose (Experimental): Participants with advanced solid tumors with or without Hippo pathway mutations will receive SW-682 tablets administered orally in continuous 28-day cycles. SW-682 dosage and frequency of administration will vary by cohort.
  Interventions: Drug: SW-682
- Part 2 Dose Expansion Cohort 1 (Experimental): Participants with mesothelioma with or without NF2 mutations will receive SW-682 tablets administered orally in continuous 28-day cycles at the recommended dose for expansion, based on Part 1 data.
  Interventions: Drug: SW-682
- Part 2 Dose Expansion Cohort 2 (Experimental): Participants with advanced solid tumors with NF2 mutations will receive SW-682 tablets administered orally in continuous 28-day cycles at the recommended dose for expansion, based on Part 1 data.
  Interventions: Drug: SW-682
- Part 2 Dose Expansion Cohort 3 (Experimental): Participants with advanced solid tumors with other Hippo pathway mutations identified during Part 1 (Phase 1a) dose escalation will receive SW-682 tablets administered orally in continuous 28-day cycles at the recommended dose for expansion, based on Part 1 data.
  Interventions: Drug: SW-682
- Part 2 Dose Expansion Cohort 4 (Experimental): Participants will receive SW-682 tablets administered orally in continuous 28-day cycles at the recommended dose for expansion, based on Part 1 data, with appropriate combination therapy, identified based on Part 1 data.
  Interventions: Drug: SW-682; Drug: Combination Therapy

INTERVENTIONS:
Drug: SW-682 — SW-682 tablet administered orally
Drug: Combination Therapy — Appropriate combination therapy
  Arms: Part 2 Dose Expansion Cohort 4

SUMMARY:
This is a first-in-human (FIH), Phase 1a/1b open-label, multicenter, dose escalation and dose expansion study of SW-682 in adult participants with metastatic or unresectable advanced solid tumors with or without Hippo pathway alterations that are refractory to, or have progressed, during or after appropriate prior systemic anticancer therapy, including chemotherapy, immunotherapy, radiation therapy or targeted therapy, or for which no treatment is available, or prior standard of care (SOC) therapy was not tolerated and for which there is no further SOC treatment available. The study includes a Part 1 (Phase 1a) dose escalation phase and a Part 2 (Phase 1b) dose expansion to optimize the dose to be used for further development. All participants will self-administer SW-682 by mouth in 28-day cycles.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed, metastatic, or unresectable solid cancer that has either not responded to or progressed during or after appropriate prior systemic anticancer therapy including chemotherapy, immunotherapy, radiation therapy, or appropriate targeted therapy, or for which there is no treatment available or prior SOC therapy was not tolerated and for which there is no further SOC treatment available
* Part 1: must have one of the following:

  * Mesothelioma with or without NF2 mutations
  * Advanced solid tumors with NF2 mutations
  * Advanced solid tumors with other Hippo pathway mutations or fusions (e.g., FAT1, LATS1/2, YAP fusions; WWTR1-CAMTA1 in EHE).
* Part 2: must have the tumor histology and oncogenic mutation or genomic aberration specific to each dose expansion cohort defined below:

  * Cohort 1: Participants with mesothelioma with or without NF2 mutations
  * Cohort 2: Participants with advanced solid tumors with NF2 mutations
  * Cohort 3: Participants with advanced solid tumors with other Hippo pathway mutations identified during Part 1 (Phase 1a) dose escalation
  * Cohort 4: SW-682 with appropriate combination therapy.
* In both parts, participants should have known oncogenic mutation identified by Next Generation Sequencing or local assay
* Must have archival tumor tissue or agree to a fresh tumor biopsy at screening
* Measurable disease per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Adequate bone marrow, kidney, hepatic, and coagulation function

Key Exclusion Criteria:

* Evidence of symptomatic CNS metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression
* Clinically significant cardiac disease or abnormal cardiac parameters
* Preexistence or inheritance of a familial renal syndrome
* Concomitant non-anti-arrhythmic medications that are known to prolong the QTc interval
* Concomitant medicines that are known strong/moderate inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) and/or CYP1A2 within 14 days or 5 half-lives before the first dose of study treatment
* Concomitant medicines that are known sensitive substrates of CYP3A4, CYP2C19, CYP2D6, CYP1A2, and/or CYP2B6 within 14 days or 5 half-lives before the first dose of study treatment
* Concomitant medicines that are known sensitive substrates of PGP, BCRP, OATP1B1, OATP1B3, OAT1, OAT3, MATE1, MATE2-K, OCT2
* Clinically significant active infection (bacterial, fungal, or viral)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Part 1 Only) | Up to 24 months
  Safety and tolerability endpoint evaluation via incidence of dose limiting toxicities (DLTs), serious adverse events (SAEs), treatment emergent adverse events (TEAE)
Maximum Tolerated Dose (Part 1 Only) | Up to 24 months
  The maximum tolerated dose (MTD) for SW-682, if any, will be based on safety and tolerability during the first 28 days of treatment in Cycle 1.
Recommended Dose for Expansion (Part 1 Only) | Up to 24 months
  The recommended dose for expansion (RDE) will be determined based on all safety, tolerability, pharmacokinetics (PK), preliminary antitumor efficacy, and other available data from Part 1 of the study.
Objective Response Rate (Part 2 Only) | Up to 24 months
  Objective response rate (ORR), defined as the proportion of participants with confirmed CR or PR using RECIST v1.1, mRECIST for mesothelioma, and/or GCIG CA-125 for ovarian cancer, as applicable, assessed by the investigator.

SECONDARY OUTCOMES:
Change in plasma and urine concentrations of SW-682 | Up to 24 months
  Plasma and urine concentrations of SW-682 and any relevant metabolite(s) will be measured to evaluate systemic exposures and renal elimination.
Objective Response Rate (Part 1 Only) | Up to 24 months
  Objective response rate (ORR), defined as the proportion of participants with confirmed CR or PR using RECIST v1.1, mRECIST for mesothelioma, and/or GCIG CA-125 for ovarian cancer, as applicable, assessed by the investigator.
Disease Control Rate | Up to 24 months
  Disease control rate (DCR), defined as the percentage of participants with CR, PR, or stable disease (SD) after starting study treatment.
Duration of Response | Up to 24 months
  Duration of response (DoR), defined as the time from response (CR + PR using RECIST v1.1, mRECIST and/or (GCIG) criteria for CA-125 response in ovarian cancer, as applicable) to disease progression and/or death, whichever occurs first.
Progression-Free Survival | Up to 24 months
  Progression-free survival (PFS), defined as the time from the date of the first administration of study treatment to the first documented disease progression per RECIST v1.1, mRECIST, and/or GCIG CA-125, as applicable, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - SpringWorks Clinical Trial Site, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - SpringWorks Clinical Trial Site, Los Angeles, California
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Knight Cancer Institute Clinical Trials, Portland, Oregon
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas